CLINICAL TRIAL: NCT03916237
Title: Utilizing a Clinical Registry and Environmental Screening Tool to Identify Children With Asthma Most Likely to Benefit From Home Assessment and Remediation
Brief Title: Registry and Screening Tool to Identify Children With Asthma Likely to Benefit From Home Assessment and Remediation
Acronym: CREST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: Cleveland Metropolitan School District (Unknown); Environmental Health Watch (Unknown); Legal Aid Society of Cleveland (Unknown)
Responsible Party: Principal Investigator, Vanessa Maier, MD, Assistant Professor & Medical Director, School Health, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB18-00771
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Asthma; Pediatric ALL; School Health Services; Registries; Medical Informatics; Home Visits; Housing Problems; Social Determinants of Health; Healthcare Disparity; Health Status Disparity
Keywords: medical legal partnership; urban health services; urban health
MeSH Terms: conditions — Asthma; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Students enrolled in the School Health Program with a diagnosis of asthma will be randomized into two groups. The first group will receive regular School Health asthma care. The second group will receive the Asthma Home Assessment Intervention. Based on results of the screening tool and home assessments, participants will be placed into one of four groups: GROUP A (no referral) GROUP B (home assessment only) GROUP C (home assessment and remediation) and GROUP D (medical legal partnership referral only) Home assessment and remediation follows Environmental Health Watch Healthy Homes model previously described. Medical Legal partnership referrals follow protocols consistent with medical legal partnerships previously prescribed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- CONTROL (No Intervention): Control group
- GROUP A no referral (Experimental): Screener does not document need for home visit or medical legal partnership referral.
  Interventions: Other: Regular School Based Health Asthma Care
- GROUP B1 home assessment only (Experimental): Screener documents need for home assessment. Home assessment does not document need for home remediation. Screener does not document need for medical legal partnership.
  Interventions: Other: Home assessment
- GROUP B2 home assessment only (Experimental): Screener documents need for home assessment. Home assessment does not document need for home remediation. Screener documents need for medical legal partnership.
  Interventions: Other: Home assessment; Other: Referral to Medical Legal Partnership
- GROUP C1 home assessment and remediation (Experimental): Screener documents need for home assessment. Home assessment documents need for home remediation. Screener does not document need for medical legal partnership.
  Interventions: Other: Home assessment; Other: Home remediation
- GROUP C2 home assessment and remediation (Experimental): Screener documents need for home assessment. Home assessment documents need for home remediation. Screener documents need for medical legal partnership.
  Interventions: Other: Home assessment; Other: Home remediation; Other: Referral to Medical Legal Partnership
- D medical legal partnership only (Experimental): Screener does not document need for home assessment. Screener does not document need for medical legal partnership.
  Interventions: Other: Referral to Medical Legal Partnership

INTERVENTIONS:
Other: Home assessment — Home assessment for environmental hazards according to protocol established by Environmental Health Watch (Healthy Home Audit https://www.ehw.org/healthy-home-audit/)
  Arms: GROUP B1 home assessment only; GROUP B2 home assessment only; GROUP C1 home assessment and remediation; GROUP C2 home assessment and remediation
Other: Home remediation — Low level home remediation according to previously established protocol (Kercsmar CM, Dearborn DG, Schluchter M, et al. Reduction in asthma morbidity in children as a result of home remediation aimed at moisture sources. Environ Health Perspect. 2006;114(10):1574-80)
  Arms: GROUP C1 home assessment and remediation; GROUP C2 home assessment and remediation
Other: Referral to Medical Legal Partnership — Medical Legal Partnership referral as described by the National Center for Medical Legal partnerships and others (Beck AF, Identifying and treating a substandard housing cluster using a medical-legal partnership. Pediatrics. 2012;130(5):831-838)
  Arms: D medical legal partnership only; GROUP B2 home assessment only; GROUP C2 home assessment and remediation
Other: Regular School Based Health Asthma Care — Regular care in the School Health Program
  Arms: GROUP A no referral

SUMMARY:
Recognizing a decline in pediatric primary care visits and immunizations rates, an increase in utilization of the emergency room and stagnating academic achievement, leaders of MetroHealth Medical Center and the Cleveland Metropolitan School District understood that an innovative delivery option would be required to meet the needs of their pediatric urban population. In the fall of 2013, with support from local and regional funders, they collaborated to open the first School Based Health Center in Cleveland. During its first year, the MetroHealth School Health Program provided primary care services to children in 98 clinical care visits. Through an emphasis on population health and care coordination, the School Health Program has grew dramatically, completing over 2,400 visits in the 2017-2018 school year at clinical sites in over 13 schools. The School Health Program has been successful in developing a care management model to improve the percentage of students who complete recommended preventive services including immunization and preventive visits. The investigators intend to apply and expand upon lessons learned to develop an effective multi component asthma care management model that includes (1) registry utilization (2) evidence based clinical care protocols (3) implementation of an Environmental Screening Tool (4) effective utilization of a Medical Legal Partnership (5) effective partnership with an environmental health justice community organization, Environmental Health Watch, for home assessment and remediation (6) utilization of a unique data sharing partnership between a large health system and school district to document health and educational outcomes.

DETAILED DESCRIPTION:
Students enrolled in the MetroHealth School Health Program (signed parental consent on file in electronic health record) and have a diagnosis of asthma on active problem list, or were seen in Emergency Department or Express Care in past 12 months for asthma related diagnosis, or have a rescue or controller inhaled medication on current medication list, will be considered for inclusion. Research staff will call families who meet inclusion criteria to discuss the study, determine interest in inclusion and obtain consent. Once enrolled baseline measures will be obtained, including level of asthma control and responses on the Environmental Screening Tool (EST) and the Community Advocacy Program Home Asthma Screening Tool (CAPHAST) (see CREST phone screening tool). Participants will then be randomized into two groups. The first group will receive regular care. The second group will receive the Asthma Home Assessment Intervention. Based on results of the screening tool and home assessments, participants will be placed into one of four groups (see CREST study design): GROUP A (no referral) GROUP B (home assessment only) GROUP C (home assessment and remediation) and GROUP D (medical legal partnership referral only) Participants randomized to regular care will be assessed for outcome measures at 3 and 6 months after randomization. Those randomized to the intervention arm will be assessed at 3 and 6 months after completion of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the MetroHealth School Health Program (signed parental consent on file in Epic electronic health record)
* Has diagnosis of asthma on active problem list OR was seen in Emergency Department or Express Care in past 12 months for asthma related diagnosis, OR has asthma related rescue or controller inhaled medication on current medication list.

Exclusion Criteria:

• Does not meet inclusion criteria.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Asthma Control Test Score | baseline and 3 and 6 months after intervention
  Score on: Asthma Control Test (for children 12 and over) or Child Asthma Control Test (for children under 12) The Asthma Control Test is used to identify asthma control with scores ranging from a minimum of 5 (poor control) to a maximum of 25 (complete control) A score of over 19 indicated well controlled asthma.

SECONDARY OUTCOMES:
Change in number of Asthma Related Emergency Department Visits | baseline and 3 and 6 months after intervention
  Self reported number of asthma related emergency department visits in past 4 months
Change in number of Asthma Related Hospitalizations | baseline and 3 and 6 months after intervention
  Self reported number of asthma related hospitalizations in past 4 months
Change in number of Asthma related Express Care or Urgent Care visits | baseline and 3 and 6 months after intervention
  Self reported number of asthma related Express Care or Urgent Care visits in past 4 months
Educational Outcome: attendance | in past 3 months
  number of absences

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Maier, MD, MPH, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No